CLINICAL TRIAL: NCT05274854
Title: A Practice Change for Patients With Severe Chronic, Clinically Unexplained Gastrointestinal Symptoms: A Randomised, Controlled Intervention to Assess Efficacy and Cost-effectiveness
Brief Title: A Practice Change for Patients With Severe Chronic, Clinically Unexplained Gastrointestinal Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Princess Alexandra Hospital, Brisbane, Australia (Other); Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APP2004495
Record Dates: First submitted 2022-02-07; First posted 2022-03-11 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Gastrointestinal Diseases; Irritable Bowel Syndrome
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — Fumigant 93

STUDY DESIGN:
Intervention Model Description: An Effectiveness-Implementation Hybrid Design with a two stage randomisation will be used to determine and compare efficacy and cost-effectiveness of different management approaches/interventions. Patients will initially receive standardised assessment of symptoms and wheat intolerance. Those patients that continue to experience symptoms will then be randomised to one of four pre-consultation interventions followed by randomisation to one of two consultation interventions conditional on their response to the initial intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preconsultation Intervention (Experimental): Pre-consultation intervention includes 4 arms ((a) standardised dietician supervised intervention, b) exercise intervention, c) internet delivered cognitive behavior therapy or d) nothing)
  Interventions: Behavioral: a)standardised dietician supervised intervention, b) exercise intervention, c) internet delivered cognitive behavior therapy or d) nothing
- Consultation Intervention (Experimental): Consultation intervention includes 2 arms (a) consultant-led outpatient clinic or b) a integrated care clinic depending on their response to the initial preconsultation intervention.
  Interventions: Behavioral: a) consultant-led outpatient clinic or b) a integrated care clinic

INTERVENTIONS:
Behavioral: a)standardised dietician supervised intervention, b) exercise intervention, c) internet delivered cognitive behavior therapy or d) nothing — Pre consultation interventions consist of one of four intervention a)standardised dietician supervised intervention, b) exercise intervention, c) internet delivered cognitive behavior therapy or d) nothing
  Arms: Preconsultation Intervention
Behavioral: a) consultant-led outpatient clinic or b) a integrated care clinic — Consultation intervention consists of one of two interventions a) consultant-led outpatient clinic or b) a integrated care clinic
  Arms: Consultation Intervention

SUMMARY:
This research project aims to test whether early interventions delivered remotely and prior to integrated care clinic appointments are effective. Patients with chronic unexplained gastrointestinal symptoms will initially undergo structured assessment of symptoms and wheat intolerance delivered remotely. Patients who continue to experience symptoms will then be randomised to a pre-consultation intervention ((a) standardised dietician supervised intervention, b) exercise intervention, c) internet delivered cognitive behavior therapy or d) nothing) followed by randomisation to the consultation intervention ((a) consultant-led outpatient clinic or b) a integrated care clinic depending on their response to the initial intervention.

DETAILED DESCRIPTION:
An Effectiveness-Implementation Hybrid Design with a two stage randomisation will be used to determine and compare efficacy and cost-effectiveness of different management approaches/interventions for patients with relevant, chronic, or relapsing gastrointestinal symptoms without concerning features and on the wait list for integrated care clinic at the Princess Alexandra Hospital. Approximately 200 patients will initially receive standardised assessment of symptoms and wheat intolerance. Those patients that continue to experience symptoms will then be randomised to a pre-consultation intervention (a) standardised dietician supervised intervention, b) exercise intervention, c) internet delivered cognitive behavior therapy or d) nothing) followed by randomisation to the consultation intervention (a) consultant-led outpatient clinic or b) an integrated care clinic conditional on their response to the initial intervention. Specific aims of the study include Aim 1: Determine efficacy (symptom improvement) and cost-effectiveness (quality adjusted life years) of a structured, digital technology enabled approach for the management of patients with severe functional gastrointestinal disorders as compared to established service models; Aim 2: Identify response-predictors for the pre-clinical dietary intervention, internet delivered cognitive behavior therapy, exercise physiology and the various clinical interventions; Aim 3: Define acceptance of consumers and staff for the new service model relative to established models of care and Aim 4. To determine the dietary patterns of people with functional gastrointestinal disorders who are presenting with symptoms necessary to access tertiary care and to further examine changes in diet after a range of interventions delivered by telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relevant, chronic, or relapsing gastrointestinal (GI) symptoms without concerning features and on the wait list for integrated care clinic (ICC) will be included in the study.
* Patients with severe symptoms as defined by a total Structured Assessment of Gastrointestinal Symptoms (SAGIS) score > 35
* Patients aged 18 years or older to 90 years old

Exclusion Criteria:

* Patients with 'alarm' signs or symptoms (significant unexplained weight loss, evidence for gastrointestinal bleeding, iron deficiency anaemia, new onset GI symptoms) will be triaged to undergo urgent clinical work-up before they can be considered for inclusion into the study
* Patients with mild or moderate symptoms (e.g. not requiring clinical work-up or who will likely spontaneously improve) will not be eligible for inclusion into the study and will be managed as clinically indicated.
* Patients with any comorbidities that would interfere with the objectives of these interventions will be managed via the routine clinical pathways.
* Patients with a prior history of any eating disorder, wait listed for bariatric surgery or have had bariatric surgery will be excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Structured Assessment of Gastrointestinal Symptoms score | Week 0
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 8
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 16
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 20
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 24
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 28
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 32
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 35
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 38
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
Structured Assessment of Gastrointestinal Symptoms score | Week 44
  Structured Assessment of Gastrointestinal Symptoms score: Assesses impact of various GI symptoms. SAGIS scores will be used to measure symptom type and symptom severity. Scores can range from 0 to 88. Higher scores indicate greater severity of symptoms
European Quality of Life Five Dimension (EQ-5D) | Week 0
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 8
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 16
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 20
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 24
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 28
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 32
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 35
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 38
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
European Quality of Life Five Dimension (EQ-5D) | Week 44
  The EQ-5D is a preference-based health related Quality of Life measure. The maximum score of 1 indicates the best health state
Cost effectiveness | Week 0
  To assess the cost-effectiveness and given the expected impact of the intervention on patient quality of life, a cost-utility analysis (CUA) will be conducted. The analysis will capture direct medical and non- medical costs including out-of-pocket expenses and indirect costs (e.g., lost productivity) based upon resources consumed using unit prices from standard costing resources. Quality-adjusted life-year (QALYs) gained will be weighted by their utility score (using the EQ-5D)
Cost effectiveness | Week 8
  To assess the cost-effectiveness and given the expected impact of the intervention on patient quality of life, a cost-utility analysis (CUA) will be conducted. The analysis will capture direct medical and non- medical costs including out-of-pocket expenses and indirect costs (e.g., lost productivity) based upon resources consumed using unit prices from standard costing resources. Quality-adjusted life-year (QALYs) gained will be weighted by their utility score (using the EQ-5D)
Cost effectiveness | Week 16
  To assess the cost-effectiveness and given the expected impact of the intervention on patient quality of life, a cost-utility analysis (CUA) will be conducted. The analysis will capture direct medical and non- medical costs including out-of-pocket expenses and indirect costs (e.g., lost productivity) based upon resources consumed using unit prices from standard costing resources. Quality-adjusted life-year (QALYs) gained will be weighted by their utility score (using the EQ-5D)
Cost effectiveness | Week 28
  To assess the cost-effectiveness and given the expected impact of the intervention on patient quality of life, a cost-utility analysis (CUA) will be conducted. The analysis will capture direct medical and non- medical costs including out-of-pocket expenses and indirect costs (e.g., lost productivity) based upon resources consumed using unit prices from standard costing resources. Quality-adjusted life-year (QALYs) gained will be weighted by their utility score (using the EQ-5D)
Cost effectiveness | Week 44
  To assess the cost-effectiveness and given the expected impact of the intervention on patient quality of life, a cost-utility analysis (CUA) will be conducted. The analysis will capture direct medical and non- medical costs including out-of-pocket expenses and indirect costs (e.g., lost productivity) based upon resources consumed using unit prices from standard costing resources. Quality-adjusted life-year (QALYs) gained will be weighted by their utility score (using the EQ-5D)

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Week 0
  Anxiety and Depression scores from the Hospital Anxiety and Depression Scale. Scores can range from 0 to 21 for each subscale of anxiety and depression, respectively. Higher scores indicate greater frequency of anxiety and depression.
Hospital Anxiety and Depression Scale | Week 16
  Anxiety and Depression scores from the Hospital Anxiety and Depression Scale. Scores can range from 0 to 21 for each subscale of anxiety and depression, respectively. Higher scores indicate greater frequency of anxiety and depression.
Hospital Anxiety and Depression Scale | Week 28
  Anxiety and Depression scores from the Hospital Anxiety and Depression Scale. Scores can range from 0 to 21 for each subscale of anxiety and depression, respectively. Higher scores indicate greater frequency of anxiety and depression.
Hospital Anxiety and Depression Scale | Week 44
  Anxiety and Depression scores from the Hospital Anxiety and Depression Scale. Scores can range from 0 to 21 for each subscale of anxiety and depression, respectively. Higher scores indicate greater frequency of anxiety and depression.
Microbiome | Week 0
  Total abundance and relative abundance of specific phyla of the microbiome
Microbiome | Week 16
  Total abundance and relative abundance of specific phyla of the microbiome
Microbiome | Week 28
  Total abundance and relative abundance of specific phyla of the microbiome
Microbiome | Week 44
  Total abundance and relative abundance of specific phyla of the microbiome
Acceptance of models of care by consumers and staff | Week 16
  For the pre-consultation and the 3- months intervention period, the consumer's net promotor score ('…I would recommend the service I received to a family member or friend yes/no..') will be determined and compared. With regard to the team providing services to the patients, all members providing care will respond to the following question in relation to specific treatment groups: '...I have been able to address the patient's problems yes/no..'
Acceptance of models of care by consumers and staff | Week 28
  For the pre-consultation and the 3- months intervention period, the consumer's net promotor score ('…I would recommend the service I received to a family member or friend yes/no..') will be determined and compared. With regard to the team providing services to the patients, all members providing care will respond to the following question in relation to specific treatment groups: '...I have been able to address the patient's problems yes/no..'

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Holtmann, MD PhD, Principal Investigator — The University of Queensland
Locations (1):
- Princess Alexandra Hospital, Woolloongabba, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
Deidentified group data will be analysed and published in medical journals